CLINICAL TRIAL: NCT02167256
Title: A Phase IIa Multi-Center Study of 18F-FDG PET, Safety, and Tolerability of AZD0530 in Mild Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Alzheimer's Therapeutic Research Institute (Other)
Responsible Party: Principal Investigator, Stephen M. Strittmatter, Professor of Neurology and Neurobiology, Yale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1404013830; 4UH3TR000967-02 (NIH)
Record Dates: First submitted 2014-06-12; First posted 2014-06-19 (Estimated); Results first posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-07

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — saracatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AZD0530 100mg daily (Experimental): Patients in the experimental group (50%) will be started on this dose. After 2 weeks, patients with a plasma drug level of <100ng/ml will receive 125mg AZD0530 daily and remain in the same experimental group as patient receiving 100mg daily.
  Interventions: Drug: AZD0530 100mg daily; Drug: AZD0530 125mg daily
- AZD0530 Placebo (Placebo Comparator): 50% of patients will receive placebo treatment for the duration of the study,
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD0530 100mg daily — All patients in experimental group (50%) will be started on 100mg AZD0530 daily
  Other Names: saracatinib
  Arms: AZD0530 100mg daily
Drug: AZD0530 125mg daily — Patients with plasma drug level <100ng/ml after 2 weeks of 100mg AZD0530 daily will receive 125mg daily of AZD0530.
  Other Names: saracatinib
  Arms: AZD0530 100mg daily
Drug: Placebo — 50% of patients will receive placebo treatment for the duration of the study.
  Other Names: saracatinib
  Arms: AZD0530 Placebo

SUMMARY:
AZD0530 is an inhibitor of Src and Abl family kinases1. It has been developed as treatment for malignancies because these kinases play a role in tumor invasion and proliferation. However, the Src family kinases (SFKs) are highly expressed in brain and have major effects on synaptic plasticity2. Moreover, the investigators have recently shown that a specific SFK, namely Fyn, is aberrantly activated by specific conformations of the Amyloid Beta (Aß) peptide from Alzheimer's disease (AD). Genetic deletion of Fyn rescues AD deficits in preclinical models. This clinical trial will test the potential benefit of AZD0530 for Alzheimer's disease modification.

ELIGIBILITY:
Inclusion Criteria

1. NIA-Alzheimer's Association core clinical criteria for probable AD
2. 18F-Florbetapir scan with evidence of elevated Aβ (based on central review)
3. Age between 55-85 (inclusive)
4. MMSE score between 18 and 26 (inclusive)
5. Stability of permitted medications for 4 weeks. In particular:

   * Stable doses of antidepressants lacking significant anticholinergic side effects (if they are not currently depressed and do not have a history of major depression within the past 1 year)
   * Cholinesterase inhibitors and memantine are allowable if stable for 12 weeks prior to screen
6. Geriatric Depression Scale less than 6 [Note: a score ≥6 on this screening scale may be permissible, if the subject is examined by a site clinician and judged not to be depressed.]
7. Study partner is available who has frequent contact with the subject (e.g., average of 10 hours per week or more), and can accompany the subject to most visits to answer questions about the subject
8. Visual and auditory acuity adequate for neuropsychological testing
9. Good general health with no disease expected to interfere with the study
10. Subject is not pregnant, lactating, or of childbearing potential (i.e., women must be two years post-menopausal or surgically sterile)
11. Modified Hachinski less than or equal to 4
12. Completed six grades of education or has a good work history
13. Must speak English or Spanish fluently

Exclusion Criteria

1. Any significant neurologic disease other than AD, such as Parkinson's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic defaults or known structural brain abnormalities
2. Screening/baseline MRI scan with evidence of infection, infarction, or other focal lesions or multiple lacunes or lacunes in a critical memory structure
3. Subjects that have any contraindications for MRI studies, including claustrophobia, the presence of metal (ferromagnetic) implants, or cardiac pacemaker
4. Major depression, bipolar disorder as described in DSM-IV within the past 1 year or psychotic features, agitation or behavioral problems within 3 months, which could lead to difficulty complying with the protocol
5. History of schizophrenia (DSM V criteria)
6. History of alcohol or substance abuse or dependence within the past 2 years (DSM V criteria)
7. Clinically significant or unstable medical condition, including uncontrolled hypertension, uncontrolled diabetes, or significant cardiac, pulmonary, renal, hepatic, endocrine, or other systemic disease in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results, or the subject's ability to participate in the study.
8. Has had a history within the last 5 years of a primary or recurrent malignant disease with the exception of non-melanoma skin cancers, resected cutaneous squamous cell carcinoma in situ, basal cell carcinoma, cervical carcinoma in situ, or in situ prostate cancer with normal prostate-specific antigen post-treatment
9. Clinically significant abnormalities in B12 or TFTs that might interfere with the study. A low B12 is exclusionary, unless follow-up labs (homocysteine (HC) and methylmalonic acid (MMA)) indicate that it is not physiologically significant.
10. Residence in skilled nursing facility.
11. Use of any excluded medication as described in study protocol
12. Current or recent participation in any procedures involving radioactive agents, including current, past, or anticipated exposure to radiation in the workplace, such that the total radiation dose exposure to the subject in a given year would exceed the limits of annual and total dose commitment set forth in the US Code of Federal Regulations (CFR) Title 21 Section 361.1. This guideline is an effective dose of 5 rem received per year.
13. Neutropenia defined as absolute neutrophils count of <1,800/microliter
14. Thrombocytopenia defined as platelet count <120x103/microliter
15. For CSF sub-study participants, a current blood clotting or bleeding disorder, or significantly abnormal PT or PTT at screening
16. Clinically significant abnormalities in screening laboratories, including:

    * Aspartate aminotransferase (AST) >1.5 times ULN
    * Alanine aminotransferase (ALT) > 1.5 times ULN
    * Total bilirubin >1.5 times ULN
    * Serum creatinine >2.0 times ULN
17. History of interstitial lung disease
18. Patients whom the PI deems to be otherwise ineligible

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2018-02-27 (Actual); Study Completion 2018-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher H van Dyck, MD, Study Director — Yale University; Paul Aisen, MD, PhD, Study Director — USC Alzheimer's Therapeutic Research Institute (ATRI)
Locations (22):
- United States (21):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - University of California, Los Angeles, Los Angeles, California
  - Yale Alzheimer's Disease Research Unit, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Wien Center for Clinical Research/Mount Sinai Medical Center, Miami Beach, Florida
  - University of South Florida - Health Byrd Alzheimer Institute, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Ann Arbor, Michigan
  - Mount Sinai School of Medicine, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - University of Pittsburgh, Alzheimer's Disease Research Center, Pittsburgh, Pennsylvania
  - Roper St. Francis Hospital, Charleston, South Carolina
  - University of Washington, Seattle, Washington
- University of British Columbia, Clinic for AD & Related Disorders, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Donohue MC, Langford O, Insel PS, van Dyck CH, Petersen RC, Craft S, Sethuraman G, Raman R, Aisen PS; Alzheimer's Disease Neuroimaging Initiative. Natural cubic splines for the analysis of Alzheimer's clinical trials. Pharm Stat. 2023 May-Jun;22(3):508-519. doi: 10.1002/pst.2285. Epub 2023 Jan 10. PMID 36627206
- [Derived] van Dyck CH, Nygaard HB, Chen K, Donohue MC, Raman R, Rissman RA, Brewer JB, Koeppe RA, Chow TW, Rafii MS, Gessert D, Choi J, Turner RS, Kaye JA, Gale SA, Reiman EM, Aisen PS, Strittmatter SM. Effect of AZD0530 on Cerebral Metabolic Decline in Alzheimer Disease: A Randomized Clinical Trial. JAMA Neurol. 2019 Oct 1;76(10):1219-1229. doi: 10.1001/jamaneurol.2019.2050. PMID 31329216

RESULTS

PARTICIPANT FLOW:
Groups:
- AZD0530 100mg/125mg Daily: AZD0530 100mg daily: All patients in experimental group (50%) were started on 100mg AZD0530 daily
  AZD0530 125mg daily: Patients with plasma drug level <100ng/ml after 2 weeks of 100mg AZD0530 daily received 125mg daily of AZD0530.
Period: Overall Study
Arm/Group | AZD0530 100mg/125mg Daily | AZD0530 Placebo
Started | 79 | 80
Completed | 58 | 70
Not Completed | 21 | 10
Not completed — Adverse Event | 13 | 6
Not completed — Withdrawal by Subject | 4 | 4
Not completed — non-compliance | 3 | 0
Not completed — Study partner unable to participate | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD0530 100mg Daily | AZD0530 Placebo | Total
Number analyzed (Participants) | 79 | 80 | 159
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 17 | 40
  >=65 years | 56 | 63 | 119
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 31 | 72
  Male | 38 | 49 | 87
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White (not Hispanic) | 74 | 68 | 142
  Black or African American | 4 | 3 | 7
  Hispanic or Latino | 1 | 6 | 7
  American Indian or Alaskan Native | 0 | 1 | 1
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 3 | 4 | 7
  United States | 76 | 76 | 152

OUTCOME MEASURES:

1. Primary Outcome: Change in Brain Glucose Uptake Measured Using 18F-FDG PET Imaging
Description: Composite measure of brain glucose uptake using F18-FDG PET in a pre-defined set of brain regions, between baseline and 12 months.
Time Frame: 12 months
Population: Number of participants is lower than total randomized participants due to a modified intent-to-treat analysis where only randomized participants who also underwent a post-baseline F18-FDG PET brain scan are included.
Measure: Mean (Standard Deviation); unit: umol/100g/min (change)
Arm/Group | AZD0530 100mg/125mg Daily | AZD0530 Placebo
Number analyzed (Participants) | 59 | 72
umol/100g/min (change) | -0.06 (0.03) | -0.05 (0.03)

2. Primary Outcome: Number of Participants With One or More Serious/Other Adverse Events Subjects With Mild AD as Assessed by Analysis of Adverse Events, Including Symptoms, and Abnormal Findings on Physical and Neurological Examinations, and Standard Labs.
Description: Assessment of any adverse effects between drug and placebo-treated subjects
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | AZD0530 100mg/125mg Daily | AZD0530 Placebo
Number analyzed (Participants) | 79 | 80
Participants
  Subjects with one or more adverse events | 73 | 68
  Subjects with one or more serious adverse events | 12 | 7

3. Secondary Outcome: The Effect of Treatment With AZD0530 on Cognitive and Behavioral Function
Description: The change in cognitive function between baseline and 12 months will be measured by the following tests:
  1. Alzheimer Disease Assessment Scale - Cognitive 11 (ADAS-cog11). Measures: Cognitive function Maximum score: 70; Minimum score: 0. Higher score equals worse cognitive function
  2. Mini-Mental State Examination (MMSE) Measures: Cognitive Function Maximum score: 30; Minimum score: 0. Higher score equal better cognitive function
  3. Alzheimer Disease Cooperative Study - Activities of Daily Living Inventory (ADCS-ADL) Measures: Ability to perform routine daily activities Maximum score: 78; Minimum score: 0. Higher score equals better ability to perform activities of daily living
  4. Clinical Dementia Rating Sum of Boxes (CDR-SO) Measures: Dementia severity Maximum score: 18; Minimum score: 0. Higher score equals more severe dementia.
Time Frame: 12 months
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | AZD0530 100mg/125mg Daily | AZD0530 Placebo
Number analyzed (Participants) | 79 | 80
Scores on a scale
  ADAS-Cog score | 7.26 (0.954) | 6.14 (0.903)
  MMSE score | -3.84 (0.575) | -3.33 (0.543)
  ADCS-ADL | -9.49 (1.263) | -7.64 (1.199)
  CDR-SO | 1.946 (0.292) | 1.468 (0.274)

4. Secondary Outcome: Percent Change in Brain Volume Before and After Treatment
Description: Change in volume of pre-defined brain regions between baseline and 12 months of treatment.
Time Frame: 12 months
Measure: Mean (Standard Error); unit: % change in volume
Arm/Group | AZD0530 100mg/125mg Daily | AZD0530 Placebo
Number analyzed (Participants) | 57 | 62
% change in volume
  Entorhinal volume change | -2.3939 (1.8138) | -3.1002 (1.7446)
  Whole brain volume change | -1.5993 (1.0569) | -1.7077 (1.0922)
  Hippocampus volume change | -0.8931 (1.8089) | -1.542 (1.9893)

5. Secondary Outcome: Cerebrospinal Fluid Levels of Total Tau, Phospho-tau (p-Tau), and Amyloid-beta 1-42 (Abeta 1-42)
Description: Measure concentration of Tau and Amyloid-beta 1-42 biomarkers in the cerebrospinal fluid between baseline and 12 months of treatment
Time Frame: 12 months
Population: Number of participants is lower than total randomized participants due to a modified intent-to-treat analysis where only randomized participants who also underwent a post-baseline cerebrospinal fluid analysis were included.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | AZD0530 100mg/125mg Daily | AZD0530 Placebo
Number analyzed (Participants) | 17 | 17
pg/ml
  CSF Total tau | 91.7448 (212.7244) | 1.2091 (131.2533)
  CSF p-Tau | 1.5837 (17.7504) | -1.9986 (13.7311)
  CSF Abeta 1-42 | -1.3383 (47.3549) | -1.3758 (43.3233)

6. Secondary Outcome: Change in Brain Glucose Uptake Measured Using 18F-FDG PET Imaging
Description: The results from the primary outcome with brain FDG-PET imaging was analyzed by ApoE genotype. Composite measure of brain glucose uptake using F18-FDG PET in a pre-defined set of brain regions, between baseline and 12 months.
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: umol/100g/min (change)
Arm/Group | AZD0530 100mg/125mg Daily | AZD0530 Placebo
Number analyzed (Participants) | 59 | 72
umol/100g/min (change)
  APOE4 carrier FDG-PET measure from baseline: number analyzed (Participants) | 37 | 47
  APOE4 carrier FDG-PET measure from baseline | -0.06 (0.03) | -0.05 (0.03)
  APOE4 non-carrier FDG-PET measure from baseline: number analyzed (Participants) | 22 | 25
  APOE4 non-carrier FDG-PET measure from baseline | -0.06 (0.03) | -0.05 (0.03)

ADVERSE EVENTS:
Time Frame: Adverse events data were collected over a period of 1 year (study duration)
Arm/Group | AZD0530 100mg/125mg Daily | AZD0530 Placebo
All-Cause Mortality (participants affected / at risk) | 1/79 | 0/80
Serious Adverse Events (participants affected / at risk) | 12/79 | 7/80
Other Adverse Events (participants affected / at risk) | 73/79 | 65/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD0530 100mg/125mg Daily (N=79) | AZD0530 Placebo (N=80)
Infections and infestations (Infections and infestations) | 4 | 0
Cardiac disorders (Cardiac disorders) | 2 | 1
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 2 | 1
Psychiatric disorders (Psychiatric disorders) | 2 | 1
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 | 0
Nervous system disorders (Nervous system disorders) | 1 | 0
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 | 0
Gastrointestinal disorders (Gastrointestinal disorders) | 1 | 1
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD0530 100mg/125mg Daily (N=79) | AZD0530 Placebo (N=80)
Gastrointestinal disorders (Gastrointestinal disorders) | 38 | 23
Psychiatric disorders (Psychiatric disorders) | 27 | 17
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 18 | 10
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 11 | 3
Investigations (Investigations) | 24 | 17
General disorders and administration site conditions (General disorders) | 15 | 9
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 13 | 7
Infections and infestations (Infections and infestations) | 28 | 24
Renal and urinary disorders (Renal and urinary disorders) | 6 | 2
Eye disorders (Eye disorders) | 5 | 1
Nervous system disorders (Nervous system disorders) | 18 | 16
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 4 | 2
Ear and labyrinth disorders (Ear and labyrinth disorders) | 3 | 1
Reproductive system and breast disorders (Reproductive system and breast disorders) | 3 | 1
Immune system disorders (Immune system disorders) | 2 | 1
Endocrine disorders (Endocrine disorders) | 1 | 0
Cardiac disorders (Cardiac disorders) | 3 | 6
Vascular disorders (Vascular disorders) | 3 | 6
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 8
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 13 | 22
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 14 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-31): https://cdn.clinicaltrials.gov/large-docs/56/NCT02167256/Prot_SAP_000.pdf